CLINICAL TRIAL: NCT06896721
Title: Effects of Nasal Administration of Dexmedetomidine on Pre-Anesthesia Sedation, Intraoperative Brain Electrical Activity, and Incidence of Agitation During Recovery in Children: a Multicenter, Large Sample, Double-Blind, Randomized Controlled Trial
Brief Title: Effects of Nasal Administration of Dexmedetomidine on Pre-anesthesia Sedation, Intraoperative Brain Electrical Activity, and Incidence of Agitation During Recovery in Children
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Fuzhou Hua (Other)
Responsible Party: Sponsor-Investigator, Fuzhou Hua, Chief Physician, Second Affiliated Hospital of Nanchang University
Organization: Second Affiliated Hospital of Nanchang University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2024-EEG-Dexmedetomidine
Record Dates: First submitted 2025-01-19; First posted 2025-03-26 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Preoperative Anxiety; Emergence Agitation
MeSH Terms: conditions — Emergence Delirium

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dexmedetomidine (Experimental)
  Interventions: Drug: Preoperative sedation with dexmedetomidine was administered nasal before surgery
- Placebo (Placebo Comparator)
  Interventions: Drug: Preoperative sedation with normal saline was administered nasal before surgery

INTERVENTIONS:
Drug: Preoperative sedation with dexmedetomidine was administered nasal before surgery — Do not drink or fast before operation. Before entering the operating room, 2 sprits of dexmedetomidine were administered intranasally (1-2ug/kg) with conventional open venous access
  Arms: Dexmedetomidine
Drug: Preoperative sedation with normal saline was administered nasal before surgery — Do not drink or fast before operation. Before entering the operating room, 2 sprits of normal saline were administered intranasally (equal volume) with conventional open venous access
  Arms: Placebo

SUMMARY:
Pre - operative anxiety and emergence agitation are common issues among pediatric patients, which have various influences on the recovery progress and prognosis of children. Nasal administration of dexmedetomidine is a convenient and non - invasive sedation technique for children. This technique can reduce the incidences of pre - operative anxiety and emergence agitation. However, there are few studies on the effect of dexmedetomidine on intraoperative electroencephalographic activities.

In view of this, the investigators elaborately designed a prospective, multi - center, large - sample - sized, double - blind, randomized - controlled clinical trial. This trial aims to provide a basis for drug selection in pediatric anesthesia, ensuring the safety and comfort of pediatric anesthesia.

The investigators plan to select 627 participants who will undergo minor surgeries under general anesthesia. Thirty minutes before the surgery, dexmedetomidine or normal saline will be administered nasally to these participants. Before the surgery, the anxiety degree and sedation score of the participants will be assessed; during the surgery, the cooperation degree of patients during anesthesia induction will be evaluated and electroencephalographic monitoring will be carried out; after the surgery, the incidence of emergence agitation, the recovery time and the analgesic score of the participants will be assessed. Throughout the whole process, the occurrence of adverse reactions of participants will be fully monitored, and the adverse reactions will be timely recorded and treated.

ELIGIBILITY:
Inclusion Criteria:

* 2≤ age ≤6 years old, gender is not limited;

  * ASA anesthesia grade I ~ II; ③ For children who intend to undergo minor surgery under general anesthesia (including but not limited to minor surgery such as ENT surgery and hernia surgery), the operation duration is expected to be no more than 2 hours; ④ Family members agree to participate in the study and voluntarily sign informed consent;

Exclusion Criteria:

* Respiratory tract infection occurs within 4 weeks before surgery;

  * Potential or other contraindications to general anesthesia;

    * There are nasal diseases, nasal bleeding, sinusitis, nasal polyps and other conditions that affect nasal absorption; ④ Heart, liver, kidney and other vital organ dysfunction or blood system diseases;

      * Allergy or intolerance to dexmedetomidine or other α2-adrenergic receptor agonists;

        * Patients with mental illness or neurological diseases;

          * Unable to complete the test, the child's guardian refused to participate; ⑧ Have participated in other clinical trials or need to participate in other clinical trials during the study period; ⑨ Other reasons that the researchers consider inappropriate to participate in this study.

Ages: 2 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 627 (Estimated)
Dates: Start 2025-03-20 (Estimated); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Success rate of preoperative sedation | 30 minutes before medication on the day of surgery
  Successful sedation was considered when participants received Ramsay sedation score ≥3 on the sedation scale 30 minutes after medication.
Incidence of emergence agitation | After extubation, patients were evaluated every 15 minutes until they were sent out of the recovery room, approximately 15 minutes to 1 hour.
  Immediately after extubation, the Pediatric Anesthesia Emergence Delirium (PAED) Scale and the 5-Point Agitation Scale for Emergence Agitation were used to assess the level of postoperative emergence agitation (EA) in the participants. Subsequent assessments were conducted every 15 minutes until the participants was transferred back to the ward. A PAED score ≥ 12 or a 5-Point Agitation Scale score > 3 could be diagnosed as emergence agitation.
Intraoperative brain electrical activity differences | 5 minutes after the end of anesthesia induction until the patient is sent out of the operating room,approximately 45 minutes to 2 hours.
  The characteristics of four kinds of brain wave α, β ,δ and θ were analyzed by professional EEG analysis software

SECONDARY OUTCOMES:
Preoperative anxiety | Before,15 minutes and 30 minutes after administration
  The modified Yale Preoperative Anxiety Scale (mYPAS) was used to quantify the anxiety level of children before and 15min and 30min after administration, respectively. There are 22 items in the scale, including activity, language, emotional expression, arousal state and dependence on parents, etc. According to the difference of each item, children's behavior is divided into grades 1~4 or 1~6, and the total score after conversion is 23.33~100 points (conversion formula: The actual score of each part = (score ÷ number of items in each part) × (100÷ number of parts)), the higher the total score, the higher the anxiety level of the child.
Degree of cooperation in anesthesia induction | After entering the operation room to before anesthesia induction,approximately 3 minutes.
  The Induction Compliance Checklist (ICC) was used to assess the child's cooperation during the anesthesia induction period after entering the operating room and before the induction of anesthesia. The checklist includes 10 negative behaviors, totaling 11 items, covering all possible reactions of the child during anesthesia induction. A score of 0 is recorded if the child exhibits no negative behaviors during induction, while a score of 1 is recorded for each negative behavior observed. The scores for each item are summed, with a maximum score of 10. A lower ICC score indicates better cooperation during the induction period. A score of 0 indicates full cooperation, 1-3 indicates moderate cooperation, and a score ≥ 4 indicates non-cooperation.
Postoperative recovery time | A period of time beginning after the withdrawal of narcotic drugs until the patient regains self-consciousness and can respond correctly to external stimuli, approximately 15 minutes to 1 hour.
  The period from the cessation of anesthetic administration until the patient regains consciousness and can respond appropriately to external stimuli.
Incidence of delayed recovery | 30 minutes after surgery.
  Participants fail to open their eyes, shake hands, or show any significant response to painful stimuli for more than 30 minutes after surgery.
Postoperative analgesia score | Immediately after recovery, the patients were re-evaluated every 15 minutes until they were sent out of the recovery room, approximately 15 minutes to 1 hour.
  Immediately after postoperative awakening, the FLACC (Face, Legs, Activity, Cry, Consolability) Pain Assessment Scale was used to evaluate the participant's pain intensity. The total score ranges from 0 to 10, with a higher score indicating a greater level of pain experienced by the participant.
Incidence of adverse reactions | Between the time the patient is sent out of the recovery room after preoperative administration, approximately 2 to 3 hours..

IPD SHARING:
Plan to Share IPD: No